CLINICAL TRIAL: NCT01428518
Title: Special Drug Use Investigation for LAMICTAL Bipolar
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115324
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with bipolar disorder: Patients with bipolar disorder prescribed lamotrigine tablets for the first time
  Interventions: Drug: Lamotrigine tablets

INTERVENTIONS:
Drug: Lamotrigine tablets — Administered according to the prescribing information in the locally approved label by the authorities.

SUMMARY:
This post-marketing surveillance study is designed to collect and assess information on safety and effectiveness of lamotrigine tablets in patients with bipolar disorder in routine clinical practice.

("LAMICTAL" is a trademark of the GlaxoSmithKline group of companies.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with bipolar disorder
* Patients treated with lamotrigine tablets for the first time

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with bipolar disorder prescribed lamotrigine tablets for the first time
Sampling Method: Probability Sample
Enrollment: 1036 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with any adverse drug reaction | 1 year

SECONDARY OUTCOMES:
Occurrence of skin disorder | 1 year
Occurrence of suicide-related event and self injurious behaviour | 1 year
Occurrence of harming others | 1 year
Occurrence of withdrawal symptoms after treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline